CLINICAL TRIAL: NCT00090610
Title: Multicenter, Randomized, Phase II Comparative Study to Compare Efficacy & Safety of Taxotere®/Carboplatin Combination Therapy vs Sequential Therapy w/ Taxotere® Then Carboplatin as Second-line Treatment of Patients w/ Relapsed, Platinum-sensitive Ovarian Cancer
Brief Title: Second-Line Treatment for Patients With Platinum-Sensitive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008381; DUKE UNIVERSITY MEDICAL CENTER (Other: Duke UMC); DUMC03
Record Dates: First submitted 2004-08-27; First posted 2004-08-31 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2012-12

CONDITIONS: Ovarian Cancer
Keywords: Relapsed ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - Combination Therapy (Experimental): Docetaxel 30mg/m2 mg IV on Days 1 and 8, in combination with carboplatin AUC 6 IV on Day 1, repeated every 21 days X 6 cycles or until disease progression
  Interventions: Drug: Docetaxel; Drug: Carboplatin
- Arm 2 - Sequential Therapy (Experimental): Docetaxel 30mg/m2 IV on Days 1 and 8, repeated every 21 days for 6 cycles until disease progression. Once subjects have completed 6 cycles of docetaxel, they receive carboplatin AUC 6 IV every 21 days for 6 cycles or until disease progression.
  Interventions: Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Docetaxel — For Arm 1: 30mg/m2 mg IV on Days 1 and 8 repeated every 21 days for six cycles until disease progression combined with carboplatin
  For Arm 2: 30mg/m2 IV on Days 1 and 8 repeated every 21 days for six cycles until disease progression followed by carboplatin
  Other Names: Taxotere
Drug: Carboplatin — Arm 1: AUC 6 IV on Days 1 and 8, repeated every 21 days for 6 cycles or until disease progression, combined with docetaxel.
  Arm 2: AUC 6 IV every 21 days for 6 cycles or until disease progression, following six cycles of treatment with docetaxel
  Other Names: Paraplatin

SUMMARY:
The purpose of this study is to compare the progression-free survival of two treatment regimens for relapsed ovarian cancer.

DETAILED DESCRIPTION:
Primary Objective

The primary objective of the study is to compare the progression-free survival of two treatment regimens:

Taxotere® 30 mg/m2 IV on Days 1 and 8, combined with carboplatin AUC 6 IV on Day 1, repeated every 21 days for 6 cycles or until disease progression. (A patient who has completed 6 cycles of treatment and who has achieved a partial response or stable disease may either continue or stop treatment at the investigator's discretion.)

Versus

Taxotere® 30 mg/m2 IV on Days 1 and 8, repeated every 21 days up to 6 cycles or until disease progression. Followed by carboplatin (AUC 6) IV every 21 days if the patient does not achieve a complete response or has disease progression on Taxotere®. A patient who has achieved a complete response on Taxotere® will be followed until the subsequent recurrence at which time she will then receive single-agent carboplatin. Carboplatin treatment will be discontinued if the patient has completed 6 cycles of treatment and has achieved a complete response or has disease progression. (A patient who has completed 6 cycles of carboplatin treatment and who has achieved a partial response or stable disease may either continue or stop treatment at the investigator's discretion.)

Secondary Objectives

The secondary objectives of the study are to compare the objective response rates (defined as a complete response plus partial response), duration of tumor response, median survival, QOL and safety in patients treated with the two regimens described above.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed epithelial ovarian cancer, peritoneal serous cancer, or tubal carcinoma.
* The patient's tumor is platinum-sensitive, which means that the patient had a complete response to front-line treatment with a platinum compound and had a treatment-free interval without clinical evidence of progressive disease for greater than 6 months.
* The patient has received one and only one prior chemotherapy regimen for the treatment of this malignancy. Prior treatment with paclitaxel and/or a platinum compound is allowed. Patients who have received consolidation treatment are allowed. Prior treatment with Taxotere® is not allowed.

  o Consolidation therapy is allowed including a different cytotoxic agent than the agent used in the front-line regimen, intraperitoneal therapy, biologic therapy, and immunotherapy.
* Patients may have received one prior regimen with a biologic therapy, either combined with cytotoxic therapy in the front-line setting, or as a single-agent for this recurrence. The biologic therapy must be discontinued at least three weeks prior to registration.
* Measurable or evaluable disease either by radiologic imaging, or physical exam, or by measurement of CA125 < 70 on two occasions at least one week apart.
* At least 3 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation portal.
* At least 3 weeks since major surgery, with full recovery. Patients who have undergone a secondary tumor debulking or cytoreductive surgery for this malignancy are excluded.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* Age > 18 years.
* Absolute neutrophil count > 1,500/mm3; platelet count > 100,000/mm3; Hemoglobin > 8.0 g/dl
* Serum bilirubin Within Normal Limits (WNL); AST or ALT and Alkaline Phosphatase must be within the range allowing for eligibility.
* If there is childbearing potential, a serum pregnancy test must be negative.
* Patients of childbearing potential must be willing to consent to using effective contraception while on treatment and for three months following the completion of treatment.
* Informed consent has been obtained.

Exclusion Criteria:

* Prior treatment with Taxotere®.
* Concurrent immunotherapy or hormonal therapy for the specific purpose of treatment for the disease. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to enrollment in order for the patient to be eligible to participate in this trial. Continuation of Hormone Replacement therapy is permitted.
* Serious concurrent medical or psychiatric illness, including serious active infection.
* Peripheral neuropathy > grade 2.
* History of other malignancy within the last 5 years, except for basal cell skin carcinoma.
* The patient is pregnant or nursing.
* Patients with a history of severe hypersensitivity reaction to cisplatin, carboplatin, mannitol, or drugs formulated with Polysorbate 80.
* Secondary debulking for this recurrence.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-10; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A Secord, MD, Study Chair — Duke University
Locations (19):
- United States (19):
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Jupiter Medical Center-Gynecology Oncology and Gynecology, Jupiter, Florida
  - Florida Hospital/Gyn/Onc Department, Orlando, Florida
  - Hematology-Onc. Assoc. of The Quad Cities, Bettendorf, Iowa
  - University of Iowa, Iowa City, Iowa
  - Franklin Square Hospital Center/MedStar Health-Section of Hematology/Oncology, Baltimore, Maryland
  - Cancer Center at Hackensack, Hackensack, New Jersey
  - Columbia University College of Physicians and Surg, New York, New York
  - Hope: A Woman's Cancer Center, Asheville, North Carolina
  - University of North Carolina/ Division of Gyn Oncology, Chapel Hill, North Carolina
  - Carolinas Medical Center/Gyn Oncology Department, Charlotte, North Carolina
  - Duke University/Division of Gynecologic Oncology, Durham, North Carolina
  - Forsyth Regional Cancer Center, Winston-Salem, North Carolina
  - Gynecologic Oncology and Surgery, Oklahoma City, Oklahoma
  - PA Hematology/Oncology Associates, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - MUSC-Div of Gyn/Oncology, Charleston, South Carolina
  - The West Cancer Clinic, Memphis, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas

REFERENCES:
- [Result] Alvarez Secord A, Berchuck A, Higgins RV, Nycum LR, Kohler MF, Puls LE, Holloway RW, Lewandowski GS, Valea FA, Havrilesky LJ. A multicenter, randomized, phase 2 clinical trial to evaluate the efficacy and safety of combination docetaxel and carboplatin and sequential therapy with docetaxel then carboplatin in patients with recurrent platinum-sensitive ovarian cancer. Cancer. 2012 Jul 1;118(13):3283-93. doi: 10.1002/cncr.26610. Epub 2011 Nov 9. PMID 22072307
- [Result] Pokrzywinski R, Secord AA, Havrilesky LJ, Puls LE, Holloway RW, Lewandowski GS, Higgins RV, Nycum LR, Kohler MF, Revicki DA. Health-related quality of life outcomes of docetaxel/carboplatin combination therapy vs. sequential therapy with docetaxel then carboplatin in patients with relapsed, platinum-sensitive ovarian cancer: results from a randomized clinical trial. Gynecol Oncol. 2011 Dec;123(3):505-10. doi: 10.1016/j.ygyno.2011.08.015. Epub 2011 Sep 25. PMID 21945310
- [Result] Havrilesky LJ, Pokrzywinski R, Revicki D, Higgins RV, Nycum LR, Kohler MF, Berchuck A, Myers ER, Secord AA. Cost-effectiveness of combination versus sequential docetaxel and carboplatin for the treatment of platinum-sensitive, recurrent ovarian cancer. Cancer. 2012 Jan 15;118(2):386-91. doi: 10.1002/cncr.26199. Epub 2011 May 19. PMID 21598242

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2004 and March 2007, 150 participants were enrolled at this multicenter study.
Pre-assignment Details: All patients were assigned
Groups:
- Arm 1: Docetaxel 30mg/m2 mg IV on Days 1 and 8, combined with carboplatin AUC 6 IV on Day 1, repeated every 21 days X 6 cycles or until disease progression
- Arm 2: Docetaxel 30mg/m2 IV on Days 1 and 8, repeated every 21 days for 6 cycles until disease progression, followed by carboplatin AUC 6 IV every 21 days for 6 cycles or until disease progression.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 75 | 75
Completed | 74 | 74
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.17) | 64.9 (10.04) | 63.9 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression in measurable disease is defined as any of the following: At least a 20% increase in the sum of the longest diameter target lesions; appearance of one or more new lesions; Death due to disease without prior objective documentation of progression; deterioration in health status attributable to the disease requiring a change in therapy without objective documentation of progression
  Progression in non-measurable disease according to CA125 levels is defined as any of the following: CA125 that begins in normal range increases to twice the upper limit of normal; CA125 level that begins elevated increases 25% over two previous samples, a 50% increase over three previous samples, or a persistent elevation over 100 U/ml for more than 2 months without a 50% decrease.
Time Frame: Every 6 months, to 18 months
Population: 1 patient in each arm was excluded. The patient in Arm 1 did not complete 1 cycle of therapy. A patient in Arm 2 withdrew from the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 74 | 74
months | 13.7 [9.9 to 16.8] | 8.4 [7.1 to 11.0]

2. Secondary Outcome: Objective Response Rate
Description: Complete response rate plus partial response rate, where: Complete response (CR) is defined as disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart and normalization of elevated CA125 in cases of ovarian cancer; Partial response (PR) for measurable disease is defined >= 30% decrease in the sum of the longest dimensions of all target measurable lesions with no unequivocal progression of non-target lesions as well as no new lesions, with documentation by two disease assessments at least four weeks apart. PR according to CA125 levels is defined as a 50% decrease in CA125 levels where two initial samples were elevated and the sample that shows the 50% is confirmed by a fourth sample 28 days after the prior sample.
  OR = CR + PR
Time Frame: Every 6 months, starting at 12 months to 24 months
Population: Same as for PFS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 74 | 74
percentage of participants | 55.4 [43.4 to 67.0] | 43.3 [31.8 to 55.3]

3. Secondary Outcome: Quality of Life
Description: Quality of Life was measured using the Trial Outcome Index (TOI) score of the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) instrument, version 4. The TOI portion of the FACT-O included questions related to Physical well-being (PWB), Social/Family well-being (FWB), and an ovarian cancer specific module (OCS). The PWB score range is from 0-28; the FWB score range is from 0-28; the OCS score range is from 0-44; this gives the TOI a score range from 0-100. (TOI = PWB + FWB + OCS)
  With these instruments, a higher score indicates better health-related quality of life.
Time Frame: Baseline performed 14 days before first dose, then every other cycle and at study termination
Population: The number of participants was based on QoL data available for Arm 1 and one patient withdrew on Arm 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 74 | 74
units on a scale
  Baseline | 76.3 (14.0) | 76.6 (16.1)
  Cycle 1 | 65.1 (21.3) | 73.3 (16.2)
  Cycle 2 | 72.7 (15.1) | 75.3 (13.6)
  Cycle 3 | 69.4 (13.5) | 75.6 (12.8)
  Cycle 4 | 70.8 (15.07) | 76.0 (13.7)
  Cycle 5 | 69.3 (14.5) | 74.0 (16.2)
  Cycle 6 | 74.3 (10.6) | 81.2 (9.7)
  End of Study | 71.4 (15.0) | 78.0 (14.8)

4. Secondary Outcome: Recurrence-Free Survival
Description: Recurrence-free survival is based on measurable disease using Kaplan-Meier estimates for the intent to treat (ITT) Population who achieved a complete response.
Time Frame: Every 6 months starting at 12 months, to 24 months
Population: Subjects who had a complete response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 13 | 9
months | 20 [13.8 to NA] — The upper bound cannot be estimated and is therefore considered unbounded. | 15.8 [10.4 to 25.4]

5. Secondary Outcome: Median Overall Survival
Time Frame: Every 6 months starting at 12 months, to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 74 | 74
months | 33.2 [32.4 to NA] — The upper bound cannot be estimated and is therefore considered unbounded. | 30.1 [29.3 to 43.9]

ADVERSE EVENTS:
Time Frame: 7-70 weeks
Description: Limited toxicity events including hematological, neurologic, hepatic, and renal toxicity were collected on the CRF. Other AEs were recorded in the patient's medical chart. The SAEs were captured from the first dose of study medication through 30 days after the last administration of study medication.
Groups:
- Arm 1: Docetaxel 30 mg/m2 intravenously (IV) on Days 1 and 8, combined with carboplatin area under the concentration versus time curve (AUC) 6 IV on Day 1, repeated every 21 days for 6 cycles or until disease progression (DP) (whichever occurred first).
- Arm2: Docetaxel 30mg/m2 IV on Days 1 and 8, repeated every 21 days for 6 cycles until disease progression, followed by carboplatin AUC 6 IV every 21 days for 6 cycles or until disease progression.
Arm/Group | Arm 1 | Arm2
Serious Adverse Events (participants affected / at risk) | 16/75 | 18/74
Other Adverse Events (participants affected / at risk) | 61/75 | 61/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=75) | Arm2 (N=74)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 7 (7)
allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
tongue edema (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Deep Thrombophlebitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarct (Cardiac disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=75) | Arm2 (N=74)
Hematologic toxicity (Blood and lymphatic system disorders) | 61 | 61
Neurotoxicity (Nervous system disorders) | 25 | 31
Hepatic (Hepatobiliary disorders) | 11 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No